CLINICAL TRIAL: NCT03680508
Title: Phase II Study of TSR-022 (Cobolimab) in Combination with TSR-042 (Dostarlimab) for the Treatment of Advanced Hepatocellular Carcinoma
Brief Title: TSR-022 (anti-TIM-3 Antibody) and TSR-042 (anti-PD-1 Antibody) in Patients with Liver Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACOBA-2017-2
Record Dates: First submitted 2018-09-18; First posted 2018-09-21 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Adult Primary Liver Cancer; Advanced Adult Primary Liver Cancer; Localized Unresectable Adult Primary Liver Cancer
Keywords: immunotherapy; PD-1; TIM-3
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TSR-022 (Cobolimab) and TSR-042 (Dostarlimab) (Experimental): Patients receive TSR-022 (cobolimab, TIM-3 binding antibody) and TSR-042 (dostarlimab, PD-1 binding antibody) via IV day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: TSR-022 and TSR-042

INTERVENTIONS:
Drug: TSR-022 and TSR-042 — immunotherapy
  Other Names: cobolimab, TIM-3 binding antibody; dostarlimab, PD-1 binding antibody

SUMMARY:
TSR-022 (cobolimab, TIM-3 binding antibody) and TSR-042 (dostarlimab, PD-1 binding antibody) may stop the growth of tumor cells by allowing the immune system to attack the cancer. This phase II trial is studying how well TSR-022 (cobolimab, TIM-3 binding antibody) and TSR-042 (dostarlimab, PD-1 binding antibody) work in combination in treating patients with locally advanced or metastatic liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the objective response rate (ORR) as determined by RECIST v1.1 of advanced hepatocellular cancer (HCC) patients treated with TSR-022 (cobolimab, TIM-3 binding antibody) and TSR-042 (dostarlimab, PD-1 binding antibody).

SECONDARY OBJECTIVES:

I. To determine the ORR as determined by the immune related Response Criteria (irRC), duration of response (DOR), time to progression (TTP), progression free survival (PFS), overall survival (OS), and alpha-fetoprotein (AFP) response of study participants.

II. To evaluate the safety profile of treated patients.

OUTLINE:

Patients receive TSR-022 (cobolimab, TIM-3 binding antibody) and TSR-042 (dostarlimab, PD-1 binding antibody) on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed hepatocellular cancer
* Barcelona Clinic Liver Cancer Stage B or C
* Cirrhosis grade of Child-Pugh class A or B7
* Subjects with HBV infection are required to be receiving effective antiviral therapy and have a viral load less than 100 IU/mL. Antiviral therapy is not required for subjects with HCV infection
* Have at least one tumor lesion that can be accurately measured according to Response Evaluation Criteria in Solid Tumor (RECIST v1.1)
* No prior systemic therapy for HCC
* Age ≥ 18 years
* ECOG performance status 0-1
* Resolved acute effects of any prior therapy to baseline or Grade ≤1 NCI CTCAE
* Have adequate hematologic function as documented by ANC ≥ 1000/μcl, platelet count ≥ 60,000/μcl, and hemoglobin ≥ 8.5 mg/dl
* Have adequate renal function as determined by a measured or calculated creatinine clearance ≥ 40 mL/min using the Cockcroft-Gault formula
* Have adequate hepatic function, as documented by ALT and AST ≤5x upper limit of normal, total bilirubin ≤3 mg/dL, and albumin ≥2.8 g/dL
* International normalized ratio (INR) or prothrombin time (PT) ≤2× ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin (PTT) is within therapeutic range of intended use of anticoagulants
* Prior local therapy, such as surgery, radioembolization, chemoembolization, or radiofrequency ablation is allowed if the index lesion(s) remains outside of the treatment field or has progressed since prior treatment
* Participants must agree to not donate blood during the study or for 90 days after the last dose of protocol therapy
* Female participant has a negative urine or serum pregnancy test within 7 days prior to taking study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 180 days after the last dose of study treatment, or is of nonchildbearing potential.
* Participant must be able to understand the study procedures and agree to participate in the study by providing written informed consent.

Exclusion Criteria:

* Participant must not be simultaneously enrolled in any interventional clinical trial
* Participant must not have had major surgery ≤ 3 weeks prior to initiating protocol therapy and participant must have recovered from any surgical effects
* Participants must not have received investigational therapy ≤4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior to initiating protocol therapy.
* Active or untreated central nervous system (CNS) and leptomeningeal metastases are excluded
* Prior therapy with any medication targeting PD-1, PD-L1, or TIM-3
* Participant must not have a known hypersensitivity to TSR-042 and TSR-022 components or excipients.
* Participants with active malignancy (other than HCC) or a prior malignancy within the past 2 years are excluded. Participants with completely resected cutaneous melanoma (early stage), basal cell carcinoma, cutaneous squamous cell carcinoma, cervical carcinoma in-situ, breast carcinoma in-situ, and localized prostate cancer are eligible
* Participant must not have serious, uncontrolled medical disorder, or nonmalignant systemic disease. Examples include, but are not limited to uncontrolled ventricular arrhythmia, uncontrolled major seizure disorder, unstable spinal cord compression, or superior vena cava syndrome.
* Unstable angina, new onset angina within last 3 months, myocardial infarction within last 6 months and current congestive heart failure New York Heart Association Class II or higher
* Known history of Human Immunodeficiency Virus (HIV) infection
* Active tuberculosis infection or other microbial infection or any active systemic infection requiring parenteral antibiotic therapy. All prior infections must have resolved following optimal therapy.
* Participant has an active autoimmune disease that has required systemic treatment in the past 2 years (.ie., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* History of idiopathic pulmonary fibrosis, interstitial lung disease, bronchial asthma, organizing pneumonia, bronchiolitis obliterans, drug-induced pneumonitis, or idiopathic pneumonitis
* History of organ transplantation including allogeneic bone marrow transplantation
* Participant has a diagnosis of immunodeficiency or has receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to initiating protocol therapy.
* Participant has received a live vaccine within 7 days of initiating protocol therapy.
* Psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant, lactating, breastfeeding, or intending to become pregnant during the study and for 180 days after the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From date of treatment until the date of best documented response, assessed up to 36 months
  Determined by RECIST v1.1 criteria

SECONDARY OUTCOMES:
Objective Response Rate (irRC) | From date of treatment until the date of best documented response, assessed up to 36 months
  Objective response as determined by the immune related Response Criteria
Duration of Response | From date of treatment until the date of progression, assessed up to 36 months
  Time from tumor response to progression
Time to progression | From date of treatment until the date of progression, assessed up to 36 months
  Time from treatment to progression of cancer
Progression free survival | From date of treatment until the date of progression or death, assessed up to 36 months
  Time from treatment to progression of cancer or death
Overall survival | From date of treatment until the date of death, assessed up to 36 months
  Time from treatment to death
AFP response | From treatment start to documentation of AFP progression, assessed up to 36 months.
  Percentage of AFP decrease from baseline to nadir
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v4.0 | From treatment until cessation of study treatment and resolution of adverse events, assessed up to 36 months
  Tabulation of adverse events, CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Jared D Acoba, MD, Principal Investigator — University of Hawaii
Locations (2):
- United States (2):
  - University of Hawaii, Honolulu, Hawaii
  - Oregon Health & Science University Knight Cancer Institute, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No